CLINICAL TRIAL: NCT01037829
Title: A Post-Marketing, Observational, Comparative Safety Study of the Novartis Pandemic Influenza A (H1N1) Vaccine(s) in Pregnant Women Versus Non-Vaccinated Pregnant Women
Brief Title: Novartis Pandemic Influenza A (H1N1) Vaccine(s) Observational Comparative Safety Study
Status: Completed | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: V111_12
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pregnancy women: Comparison of pregnancy outcomes between (Novartis) H1N1 vaccinated women and (Novartis) H1N1 unvaccinated women.
  Interventions: Other: Non-intervention observational study

INTERVENTIONS:
Other: Non-intervention observational study — Non-intervention observational study

SUMMARY:
The primary objective of this observational, comparative safety study is to evaluate the safety of the Novartis Pandemic Influenza A (H1N1) vaccine in pregnant women and their off spring, followed for up to 3 months of age as compared to pregnant women who have not received the Novartis Pandemic Influenza A (H1N1) vaccine. This study will be conducted at investigative sites within the Netherlands, Italy, and Argentina.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant OR was pregnant following the introduction of the Novartis Pandemic Influenza A (H1N1) vaccine in the country of interest and have already experienced a pregnancy outcome
* Consents to participate in the study

Exclusion Criteria:

* Is not currently pregnant OR was not pregnant at the time of or after the introduction of the Novartis Pandemic Influenza A (H1N1) vaccine in the country of interest
* Does not consent to participate in the study
* Has received a non-Novartis pandemic influenza vaccinee

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 4529 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Normal live-born delivery | 3 months follow-up on all live births
Spontaneous and elective abortions | 3 months follow-up on all live births
Congenital malformations | 3 months follow-up on all live births
Pre-term birth (prematurity) | 3 months follow-up on all live births
Low birth weight | 3 months follow-up on all live births
Neonatal mortality | 3 months follow-up on all live births

SECONDARY OUTCOMES:
Maternal complications of gestational diabetes, preeclampsia, maternal death | During pregnancy and post delivery

CONTACTS AND LOCATIONS:
Locations (16):
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Villa Nueva
- Italy (12):
  - Bari
  - Cagliari
  - Como
  - Milan
  - Monza
  - Prato
  - Roma
  - Rome
  - Siena
  - Trieste
  - Udine
  - Vicenza
- Podiumweg, Ilsselstein, Netherlands